CLINICAL TRIAL: NCT02932592
Title: evAluation of Glycemic RangE During acutE Coronary syndroME in Nondiabetic paTients
Brief Title: evAluation of Glycemic RangE During acutE Coronary syndroME in Nondiabetic paTients (AGREEMENT)
Acronym: AGREEMENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, MD, PhD, FESC, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20160000072
Record Dates: First submitted 2016-09-30; First posted 2016-10-13 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: CGMS
Masking Description: CGMS
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dysglycemic group (Experimental): Patients with dysglycemia (not diabetic patients) will be undergone a monitoring of blood glucose with a device till the discharge of the patient.
  Then, an oral glucose tolerance test (OGTT) will be done to categorize the patient as having impaired fasting glucose (IFG) or impaired glucose tolerance (IGT), or diabetes mellitus.
  Interventions: Device: Continuous Glucose Monitoring System (i Pro 2 - Medtronic)

INTERVENTIONS:
Device: Continuous Glucose Monitoring System (i Pro 2 - Medtronic) — This device can register blood glucose values and excursions. This device consists of a needle (applied in subcutaneous way) and of a recording device.

SUMMARY:
To evaluate the glycemic variations during acute coronary syndrome in non-diabetic patients (euglycemic, or with impaired fasting glucose, or with impaired glucose tolerance)

DETAILED DESCRIPTION:
All nondiabetic patients with dysglycemia (fasting plasma glucose between 100 and 125 mg/dl) will be monitored with a device (Continuous Glucose Monitoring System) and all these patients will be undergone an oral glucose tolerance test after the discharge from this Unit.

ELIGIBILITY:
Inclusion Criteria:

* nondiabetic patients
* acute coronary syndrome

Exclusion Criteria:

* diabetic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Glycemic status | 15 days
  Patients with dysglycemia (not diabetic patients) will be undergone a monitoring of blood glucose with a device till the discharge of the patient.
  Then, an oral glucose tolerance test (OGTT) will be done to categorize the patient as having impaired fasting glucose (IFG) or impaired glucose tolerance (IGT), or diabetes mellitus.

SECONDARY OUTCOMES:
Lipid profile | 15 days
  Total cholesterol
Lipid profile | 15 days
  HDL-cholesterol
Lipid profile | 15 days
  Triglycerides
Lipid profile | 15 days
  Lipoprotein (a)
Endothelial damage | 15 days
  sICAM-1
Endothelial damage | 15 days
  sVCAM-1
Inflammation parameters | 15 days
  sRAGE
Inflammation parameters | 15 days
  sCD40L
Inflammation parameters | 15 days
  MPO
Inflammation parameters | 15 days
  hs-CRP
Inflammation parameters | 15 days
  IL-6
Inflammation parameters | 15 days
  TNF-alfa
Heart damage | 15 days
  CPK
Heart damage | 15 days
  I troponin

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, PhD, FESC, Principal Investigator — University of Pavia
Locations (1):
- Giuseppe Derosa, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No